CLINICAL TRIAL: NCT03219502
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) to Treat Oxaliplatin-Induced Neuropathy
Brief Title: rTMS in Improving Neuropathy in Patients With Stage I-IV Cancer Who Have Received Oxaliplatin Chemotherapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-1134; NCI-2018-02093 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-1134 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Malignant Neoplasm; Neuropathy
MeSH Terms: conditions — Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (rTMS) (Experimental): Patients undergo rTMS over 30 minutes for 10 sessions over 10 business days.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Repetitive Transcranial Magnetic Stimulation
- Group II (sham rTMS) (Sham Comparator): Patients undergo sham rTMS over 30 minutes for 10 sessions over 10 business days.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Sham Intervention
- Group III (standard of care) (Active Comparator): Patients receive standard of care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Group III (standard of care)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Repetitive Transcranial Magnetic Stimulation — Undergo rTMS
  Other Names: rTMS
  Arms: Group I (rTMS)
Procedure: Sham Intervention — Undergo sham rTMS
  Arms: Group II (sham rTMS)

SUMMARY:
This trial studies how well repetitive transcranial magnetic stimulation (rTMS) works in improving neuropathy due to oxaliplatin chemotherapy in patients with stage I-IV cancer. rTMS is designed to change brain activity by introducing small magnetic impulses to the scalp that encourage the brain to change its activity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the effects of the repetitive transcranial magnetic stimulation (rTMS) training program on perceptions of chemotherapy-induced peripheral neuropathy (CIPN) versus placebo (PC) and wait-list control groups (WLC).

SECONDARY OBJECTIVES:

I. Explore changes in cortical activity: Electroencephalography (EEG) brain maps (low resolution electromagnetic tomography) will be assessed over time and compared between groups.

II. Determine if rTMS improves other aspects of CIPN, quality of life (QOL), and mental health (MH) compared to PC and WLC.

III. Explore moderators/mediators of the intervention by examining the extent to which changes in EEG patterns mediate the effects of the intervention and the extent to which there are interaction effects of the intervention and each of the baseline brain regions.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I: Patients undergo rTMS over 30 minutes for 10 sessions over 10 business days.

GROUP II: Patients undergo sham rTMS over 30 minutes for 10 sessions over 10 business days.

GROUP III: Patients receive standard of care.

After completion of study, patients are followed up within 1 week and at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage I-IV cancers who received oxaliplatin chemotherapy
* Understand and read English, sign a written informed consent, and be willing to follow protocol requirements
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Grade 2 or higher neuropathic symptoms according to the National Cancer Institute's 4 point grading scale
* Neuropathic symptoms must be related to chemotherapy (in the opinion of the treating physician)
* Patients must have neuropathic symptoms for a minimum of 3 months
* No plans to change the type of pain medication (if a patient is on pain medication)
* Willing to come to MD Anderson for the therapy sessions

Exclusion Criteria:

* Patients who are taking any antipsychotic medications
* Patients who have evidence of brain metastases or any with any active central nervous system (CNS) disease at their time of entry into the trial
* Patients who have ever been diagnosed with bipolar disorder or schizophrenia
* Patients who have a history of head injury, focal brain lesions, or known seizure activity
* Patients who are withdrawing from drugs
* Patients with intracranial implants or a cardiac pacemaker or any device that is not considered magnetic resonance imaging (MRI) safe. Colorectal patients are sometimes prescribed Tramadol to help control the symptoms of CIPN. Tramadol does lower the seizure threshold, however these patients will be considered eligible for the study if they discontinue the drug 48 hours before the baseline and do not use it during the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in perceptions of chemotherapy-induced peripheral neuropathy (CIPN) | Baseline up to 1 month
  Differences between repetitive transcranial magnetic stimulation (rTMS) and placebo (PC) and between rTMS and wait-list control (WLC) will be assessed by Pain Quality Assessment Scale (PQAS). Will conduct two-sample t-tests, subtracting post-intervention scores from pre-intervention scores at each post-intervention time point.
  The Pain Quality Assessment Scale (PQAS) is a 20-item measure developed to quantify quality and intensity of neuropathic pain. It was derived from the Neuropathic Pain Scale and includes symptom descriptors common to people with neuropathic symptoms.[44] Our primary outcome will be the 'unpleasantness subscale'.

SECONDARY OUTCOMES:
Change in cortical activity | Baseline up to 1 month
  Will include pre, interim, and post comparisons of the electroencephalography (EEG), via low resolution electromagnetic tomography (LORETA) imaging software, on an individual basis. These analyses will include global differences in cortical activation as well as site-specific dominant frequencies for each patient.
Change in perception of improvement in CIPN as assessed by Patients' Global Impression of Change (PGIC) questionnaire | Baseline up to 1 month
  Will use data across the set of post-intervention assessment points. Will conduct two-sample t-tests, subtracting post-intervention scores from pre-intervention scores at each post-intervention time point.
  The Patients' Global Impression of Change (PGIC) will measure clinically important change from the patient's perspective. Patients report symptoms on a range from "very much worse" to "very much improved".
Change in perception of improvement in CIPN as assessed by Edmonton Symptom Assessment System (ESAS) questionnaire | Baseline up to 1 month
  Will use data across the set of post-intervention assessment points. Will conduct two-sample t-tests, subtracting post-intervention scores from pre-intervention scores at each post-intervention time point.
  The Edmonton Symptom Assessment System (ESAS) is a validated tool to assess 12 major symptoms (rated 0-10) that are common in cancer patients during the 24 hours preceding its administration. The symptoms assessed are pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, insomnia, well-being, financial distress, and spiritual distress.
Change in perception of improvement in CIPN as assessed by Brief Pain Inventory-short form (BPI) questionnaire | Baseline up to 1 month
  Will use data across the set of post-intervention assessment points. Will conduct two-sample t-tests, subtracting post-intervention scores from pre-intervention scores at each post-intervention time point.
  The Brief Pain Inventory-short form (BPI) is a validated, widely used, questionnaire that will assess severity and impact of pain. We will prioritize assessment of the 'worst pain' subscale, and 'interference' subscale as they have been used to assess pain in other pain trials.
Change in perception of improvement in CIPN as assessed by Pain Vigilance and Awareness Questionnaire (PVAQ) | Baseline up to 1 month
  Will use data across the set of post-intervention assessment points. Will conduct two-sample t-tests, subtracting post-intervention scores from pre-intervention scores at each post-intervention time point.
  The Pain Vigilance and Awareness Questionnaire (PVAQ) will assess attention to pain in terms of awareness, consciousness, vigilance, and observation of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Prinsloo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org